CLINICAL TRIAL: NCT02135510
Title: MEtoclopramide, DExamethasone or Axoli (Palonoseton) for the Prevention of Delayed Chemotherapy-induced Nausea and Vomiting in Moderately Emetogenic Non-AC-based Chemotherapy: the MEDEA-trial
Brief Title: MEtoclopramide, DExamethasone or Axoli to Prevent or Delay Chemotherapy-induced Nausea and Vomiting in Moderately Emetogenic Non-AC-based Chemotherapy
Acronym: MEDEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Noordwest Ziekenhuisgroep (Other); Rijnstate (Unknown); Tergooiziekenhuizen locatie Hilversum (Unknown); Ziekenhuis Amstelland (Other)
Responsible Party: Principal Investigator, H.M.W. Verheul, Head Department Medical Oncology, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/366
Record Dates: First submitted 2014-05-01; First posted 2014-05-12 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Metoclopramide; Palonosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- metoclopramide (Active Comparator)
  Interventions: Drug: metoclopramide
- dexamethason (Active Comparator)
  Interventions: Drug: dexamethason
- palonosetron (Active Comparator)
  Interventions: Drug: palonosetron

INTERVENTIONS:
Drug: metoclopramide
  Arms: metoclopramide
Drug: dexamethason
  Arms: dexamethason
Drug: palonosetron
  Arms: palonosetron

SUMMARY:
In this phase III non-inferiority trial, the aim is to evaluate whether metoclopramide and palonosetron prophylactic antemetic treatment are non-inferior to dexamethasone with regard to its efficacy to prevent delayed chemotherapy-induced nausea and vomiting (CINV) induced by non- anthracyclines plus cyclophosphamide (AC) based moderately emetogenic chemotherapy (MEC).

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with histologically or cytologically confirmed solid cancer
* Starting with first cycle of chemotherapy of moderate emetogenic risk, which does not include a combination of anthracycline plus cyclophosphamide
* Age ≥ 18
* WHO ≤ 1
* Patient is able to understand and speak Dutch

Exclusion Criteria:

* Patient with nausea and/or vomiting in 48 hours before start of chemotherapy treatment
* Patient submitted to concomitant radiotherapy or submitted to radiotherapy 15 days before start of chemotherapy or planned to receive radiotherapy during 8 days after administration of chemotherapy
* Patient with concomitant severe comorbidy, such as: o Intestinal obstruction o Active peptic ulcer o Hypercalcemia o Uncontrolled diabetes mellitus o Pheochromocytoma o Tardive dyskinesia o Epilepsia o Active infective diseases o Brain - or leptomeningeal metastases o Psychiatrical disorders o Parkinsonism
* Current use of corticosteroids (similar to prednisone ≥ 10 milligrams per day)
* Current alcohol abuse
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2013-06; Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
efficacy | 24 to 160 hours
  Primary efficacy endpoint: the proportion of patients reporting complete response during the overall 24 to 160 hours after initiation of the first cycle of moderately emetogenic chemotherapeutic (MEC). Complete response is defined as no vomiting and nausea and no use of rescue medication. A diary will be used to document the date and time of any emetic episodes and use of rescue medication, as well as daily nausea ratings.
tolerability | 24 to 160 hours
  Primary tolerability endpoint: the proportion of patients with minimal or no antiemetic therapy-related side effects according to the Dexamethasone Symptom Questionnaire (DSQ) questionnaire, the Abnormal Involuntary Movement Scale (AIMS) and Aprepitant questionnaire during the first cycle of moderately emetogenic chemotherapeutic (MEC).
cost-effectiveness | 24 to 160 hours
  Primary cost-effectiveness endpoint: total antiemetic medication costs per treatment regimen during the first cycle of Moderately Emetogenic Chemotherapy (MEC). A diary will be used to document the use of antiemetics and rescue medication. Total medication costs will be calculated from this.

CONTACTS AND LOCATIONS:
Locations (7):
- Netherlands (7):
  - Medisch Centrum Alkmaar, Alkmaar, North Holland
  - Ziekenhuis Amstelland, Amstelveen, North Holland
  - Gemini Ziekenhuis, Den Helder, North Holland
  - Tergooiziekenhuizen, Hilversum, North Holland
  - Waterland Ziekenhuis, Purmerend, North Holland
  - De Heel - Zaans Medisch Centrum, Zaandam, North Holland
  - Rijnstate, Arnhem

REFERENCES:
- [Derived] van der Vorst MJDL, Toffoli EC, Beusink M, van Linde ME, van Voorthuizen T, Brouwer S, van Zweeden AA, Vrijaldenhoven S, Berends JC, Berkhof J, Verheul HMW. Metoclopramide, Dexamethasone, or Palonosetron for Prevention of Delayed Chemotherapy-Induced Nausea and Vomiting After Moderately Emetogenic Chemotherapy (MEDEA): A Randomized, Phase III, Noninferiority Trial. Oncologist. 2021 Jan;26(1):e173-e181. doi: 10.1634/theoncologist.2020-0305. Epub 2020 Aug 21. PMID 32735029